CLINICAL TRIAL: NCT06575400
Title: A Phase 1, Randomised, Single-blind, Placebo-controlled Trial to Assess Safety, Tolerability, and Pharmacokinetics of Single and Multiple Rising Subcutaneous Doses of BI 3804379 in Healthy Male and Female Subjects
Brief Title: A Study to Test How Well Different Doses of BI 3804379 Are Tolerated by Healthy People
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1524-0001; 2024-513549-36-00 (Registry Identifier: CTIS); U1111-1306-8874 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-08-27; First posted 2024-08-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SRD Part: BI 3804379 (Experimental): SRD= Single rising dose
  Interventions: Drug: BI 3804379
- SRD Part: Placebo matching BI 3804379 (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3804379
- MRD Part: BI 3804379 (Experimental): MRD=Multiple rising dose.
  Interventions: Drug: BI 3804379
- MRD Part: Placebo matching BI 3804379 (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3804379

INTERVENTIONS:
Drug: BI 3804379 — BI 3804379
  Arms: MRD Part: BI 3804379; SRD Part: BI 3804379
Drug: Placebo matching BI 3804379 — Placebo matching BI 3804379
  Arms: MRD Part: Placebo matching BI 3804379; SRD Part: Placebo matching BI 3804379

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PKs) of BI 3804379 in healthy male and female subjects following administration of single rising doses and administration of multiple rising doses.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male or female (of non-child-bearing potential) subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), respiratory rate (RR), temperature (TEMP)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 65 years (inclusive)
3. Body mass index (BMI) of 18.5 to 30.0 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH Harmonized Guideline for Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial Further inclusion criteria apply

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
2. Repeated measurement of systolic BP outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic BP outside the range of 45 to 90 mmHg, or PR outside the range of 45 to 100 beats per minute (bpm).
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
4. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders that the investigator considers to be of clinical relevance.

Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
SRD part and MRD part: Occurrence of any treatment-emergent adverse event (AE) assessed as drug-related by the investigator | Up to Day 84 for SRD part and up to Day 235 for MRD part.

SECONDARY OUTCOMES:
SRD part: AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to Day 84.
SRD part: Cmax (maximum measured concentration of the analyte in plasma) | Up to Day 84.
MRD part: AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to Day 235.
MRD part: Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to Day 235.

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com